CLINICAL TRIAL: NCT01295307
Title: Clofarabine Salvage Therapy in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Clofarabine Salvage Therapy in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Acronym: BRIDGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Schetelig Johannes, PD Dr. med. Johannes Schetelig, Technische Universität Dresden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUD-BRIDGE-046; 2010-022584-35 (EudraCT Number)
Record Dates: First submitted 2011-02-04; First posted 2011-02-14 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; relapsed; refractory; Relapsed or refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Clofarabine

ARMS (1):
- Single Arm (Experimental): Induction therapy with clofarabine/cytarabine. Post-remission therapy with either allogeneic HCT after conditioning with clofarabine/melphalan if a donor is available, or clofarabine/cytarabine if no donor is available
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — Induction and consolidation therapy / conditioning therapy with Clofarabine

SUMMARY:
In relapsed or refractory AML allogeneic HCT is considered to be the only treatment by which long-term disease-free survival can be achieved. Despite this favorable prospect, even in younger patients with relapsed AML only about 40% of the patients reach allogeneic HCT. A number of factors contribute to this low rate of transplantation, among them moderate activity of the salvage regimens and accumulating toxicities which prevent from transplantation; Prospective clinical trials in this indication usually focus either on the rate of CR achieved after a defined number of cycles of salvage therapy or on transplantation modalities. The consequent integration of salvage therapy into a transplant strategy accounting for the time-dependent process of donor search has not been studied so far.

The objective of this study is to evaluate the safety and efficacy of clofarabine salvage therapy prior to allogeneic HCT.

DETAILED DESCRIPTION:
All patients are scheduled for at least one cycle of induction therapy with CLARA. CLARA contains clofarabine 40 mg/m2 (1 hr infusion) days 1-5 followed 3 hours after the end of infusion by intermediate dose cytarabine 1 g/m2 (2 hrs infusion) days 1-5. Patients with moderate early response (reduced marrow blast count but ≥10% at day 15) or patients with progressive disease during delayed hematologic recovery (beyond day 42) may receive re-induction therapy similar to the first cycle induction therapy.

Study treatment comprises up to two cycles of induction therapy and one to two cycles of consolidation chemotherapy for patients without a donor. Consolidation therapy is reduced by 25% and consists of clofarabine 40 mg/m2 (1 hr infusion) days 1-4 followed 3 hours after the end of infusion by intermediate dose cytarabine 1 g/m2 (2 hrs infusion) days 1-4.

Patients for whom a donor can be identified may proceed to allogeneic HCT after CLARA I adopting the concept of allogeneic HCT in aplasia. Patients for whom donor search is more time consuming should proceed to allogeneic HCT once a donor has been identified.

Patients who have achieved a response after the last cycle of CLARA will receive clofarabine as part of the conditioning regimen. Clofarabine and melphalan may only be given as conditioning therapy to patients with HLA-compatible donors with a maximum of one mismatch refering to the HLA-loci A, -B, -C and -DRB1. Conditioning therapy then contains clofarabine 30 mg/m2 (1 hr IV infusion) days -6 to -3 and melphalan 140 mg/m2 (1 hour IV infusion) on day -2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML according to WHO criteria.
* Untreated relapse or refractory disease after a minimum of one standard induction therapy. Treatment of relapse with leukocyte-apheresis or up to 5 days with low dose cytarabine or hydroxyurea is allowed.

  * Refractory disease is defined as ≥5% blasts after the second cycle of induction therapy or no reduction in marrow blasts at early treatment assessment (day +15) after the first cycle of induction therapy.
  * Relapse is defined as an increase in bone marrow blast count ≥5%, re-appearance of blasts in the peripheral blood or extramedullary disease.
* Age above 40 years.
* Have adequate renal and hepatic functions as indicated by the following laboratory values:

  * Serum creatinine <=1.0 mg/dL; if serum creatinine >1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be >60 mL/min/1.73 m2 (see reference below*)
  * Serum bilirubin <=1.5× upper limit of normal (ULN)
  * Aspartate transaminase (AST)/alanine transaminase (ALT) <=2.5× ULN
  * Alkaline phosphatase <=2.5× ULN
* Eligibility for intensive chemotherapy
* Patient needs to be capable to understand the clinical trial as an investigational approach to bridge the time to potential allogeneic HCT, potential risks and benefits of the study.
* Signed written informed consent.
* Female patients of childbearing potential must have a negative serum
* Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.

Exclusion Criteria:

* For refractory disease, more than two prior induction chemotherapies or more than one prior salvage chemotherapy containing high-dose cytarabine (cumulative dose of cytarabine ≥ 5 g/m2).
* Second or higher relapse. Patients who received hypomethylating agents like azacytidine or decitabine as a treatment of first relapse, respond and relapse later on may be included.
* Acute promyelocytic leukemia with t(15;17)(q22;q12) molecular detection or (PML/RARα).
* Central nervous system involvement (i.e. WBC ≥ 5/µL in cerebrospinal fluid with blasts present on cytospin).
* Prior allogeneic HCT
* Autologous transplantation within 100 days prior to start of study treatment
* Use of investigational agents or anticancer therapy within 10 days before study entry with the exception of hydroxyurea or low-dose cytarabine.
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo transplantation.
* Patients with known refractoriness to platelet support.
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Pregnant or lactating patients.
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2011-03; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Rate of treatment success | To be evaluated 42 days after start of last cycle of chemotherapy containing clofarabine
  Treatment success is defined as a complete remission (CR, CRi or CRchim) at final response assessment after having completed the study treatment. CR and CRi are defined according to standard criteria (ELN). Complete remission by chimerism (CR chim) is defined as a >95% overall donor chimerism assessed by STR-PCR in bone marrow and absence of extramedullary disease together with an absolute neutrophil count >0.5 /nL (500/μL).

SECONDARY OUTCOMES:
Rate of transplantation | see evaluation of primary endpoint
  Rate of patients who finally proceeded to allogeneic HCT after bridging therapy with Clofarabine
Adverse drug reactions | see evaluation of primary endpoint
  Rate of adverse drug reactions.
Treatment failure | see evaluation of primary endpoint
  Cause specific analysis of treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Schetelig, MD, Principal Investigator — Universitätsklinikum Dresden, Med. Klinik und Poliklinik I, Study Alliance Leukemia
Locations (10):
- Germany (10):
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Klinikum Chemnitz gGmbH, Chemnitz
  - University Hospital Carl Gustav Carus, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - Klinikum der J. W. Goethe-Universität, Frankfurt am Main
  - Klinikum Mannheim GmbH, Mannheim
  - Universitätsklinikum Münster, Münster
  - Klinikum Nürnberg Nord, Nuremberg
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Würzburg, Würzburg

REFERENCES:
- [Result] Middeke JM, Herbst R, Parmentier S, Bug G, Hanel M, Stuhler G, Schafer-Eckart K, Rosler W, Klein S, Bethge W, Bitz U, Buttner B, Knoth H, Alakel N, Schaich M, Morgner A, Kramer M, Sockel K, von Bonin M, Stolzel F, Platzbecker U, Rollig C, Thiede C, Ehninger G, Bornhauser M, Schetelig J. Clofarabine salvage therapy before allogeneic hematopoietic stem cell transplantation in patients with relapsed or refractory AML: results of the BRIDGE trial. Leukemia. 2016 Feb;30(2):261-7. doi: 10.1038/leu.2015.226. Epub 2015 Aug 18. PMID 26283567
- See also: Download PDF — http://www.nature.com/leu/journal/vaop/ncurrent/full/leu2015226a.html